CLINICAL TRIAL: NCT02041598
Title: DREAM Project Community Health Worker Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-0510; P60MD000538 (NIH); U48DP001904 (NIH)
Record Dates: First submitted 2014-01-16; First posted 2014-01-22 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full CHW Intervention (Experimental): 5 monthly group educational sessions, 2 1v1 Visits with CHW, Phone Calls as Needed
  Interventions: Other: CHW Intervention
- Control: Intro to Diabetes Session Only (No Intervention): One-time, Introduction to Diabetes educational session only

INTERVENTIONS:
Other: CHW Intervention — 5 group educational sessions, 2 1v1 Visits with a CHW, Phone Calls as needed during 6-month study period
  Arms: Full CHW Intervention

SUMMARY:
The DREAM (Diabetes Research, Education, and Action for Minorities) Project is a Community Health Worker (CHW) intervention to improve diabetic management and control among Bangladeshis with diabetes in New York City (NYC).

DETAILED DESCRIPTION:
The DREAM (Diabetes Research, Education, and Action for Minorities) Project is a Community Health Worker (CHW) intervention to improve diabetic management and control among Bangladeshis with diabetes in New York City (NYC). For a two-arm, randomized controlled trial (RCT), investigators will recruit a sample of 256 participants, all of whom are 1) of Bangladeshi descent, 2) residing in NYC, 3) diagnosed with Type 2 diabetes mellitus (T2DM) and a recent Hemoglobin A1c (HbA1c) of ≥ 6.5, and 4) between the ages of 21-85. The treatment group receives a six-month CHW-led intervention consisting of five monthly group educational sessions, two one-on-one visits, and follow-up phone calls as needed from a CHW. The control group receives an introductory educational session only. Primary and secondary outcomes include clinical and behavioral measures, such as HbA1c and weight change, access to and utilization of care (i.e. appointment keeping and use of specialty care), and knowledge and practice of physical activity and healthful eating. Additionally, information regarding CHW characteristics, the processes and mechanisms for influencing healthful behavior change, and fidelity of the intervention are collected. Outcomes are measured at Baseline, 3-Months, 6-Months for both groups, and at 12-Months for the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* confirmed clinical diagnosis of T2DM with a Hemoglobin A1c (HbA1c) of ≥ 6.5%; and
* male or female between the ages of 21-85 years old; and
* willingness to be randomized to either treatment or control groups.

Exclusion Criteria:

* is or was on renal dialysis;
* experiencing an acute or terminal illness or serious mental illness;
* had a history of recent coronary event within the last 3 months of recruitment;
* is pregnant at the time of recruitment;
* experienced other severe medical conditions that might preclude participation;
* has poor short-term prognosis (expected death in <2 years); or
* is participating in another research study.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-25 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Hemoglobin A1c at 6-Months | Baseline, 6-Months
  Change in Baseline HbA1c at 6-Months

SECONDARY OUTCOMES:
Change in Baseline Perceived Social Support at 6-Months | Baseline, 6-Months
  Assessed using scale items on questionnaire instrument administered during semi-structured interview at each timepoint
Change in Baseline Perceived Benefits & Barriers at 6-Months | Baseline, 6-Months
  Assessed using scale items on questionnaire instrument administered during semi-structured interview at each timepoint
Change in Baseline Self-Efficacy at 6-Months | Baseline, 6-Months
  Assessed using scale items on questionnaire instrument administered during semi-structured interview at each timepoint
Change in Baseline Access to / Utilization of healthcare at 6-Months | Baseline, 6-Months
  Assessed using scale items on questionnaire instrument administered during semi-structured interview at each timepoint
Change in Baseline Diabetic Management Practices & Knowledge at 6-Months | Baseline, 6-Months
  Assessed using scale items on questionnaire instrument administered during semi-structured interview at each timepoint
Change in Baseline Engagement in Physical Activity & Healthy eating at 6-Months | Baseline, 6-Months
  Assessed using scale items on questionnaire instrument administered during semi-structured interview at each timepoint
Change in Baseline Lipid Profile at 6-Months | Baseline, 6-Months
  HDL, LDL, Triglycerides, Total Cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, PhD, Principal Investigator — New York University School of Medicine, Department of Population Health
Locations (1):
- New York University School of Medicine, Dept of Population Health, New York, New York, United States

REFERENCES:
- [Background] Islam NS, Wyatt LC, Patel SD, Shapiro E, Tandon SD, Mukherji BR, Tanner M, Rey MJ, Trinh-Shevrin C. Evaluation of a community health worker pilot intervention to improve diabetes management in Bangladeshi immigrants with type 2 diabetes in New York City. Diabetes Educ. 2013 Jul-Aug;39(4):478-93. doi: 10.1177/0145721713491438. Epub 2013 Jun 7. PMID 23749774
- [Derived] Wyatt LC, Katigbak C, Riley L, Zanowiak JM, Ursua R, Kwon SC, Trinh-Shevrin C, Islam NS. Promoting Physical Activity Among Immigrant Asian Americans: Results from Four Community Health Worker Studies. J Immigr Minor Health. 2023 Apr;25(2):291-305. doi: 10.1007/s10903-022-01411-y. Epub 2022 Oct 23. PMID 36273386
- [Derived] Islam N, Riley L, Wyatt L, Tandon SD, Tanner M, Mukherji-Ratnam R, Rey M, Trinh-Shevrin C. Protocol for the DREAM Project (Diabetes Research, Education, and Action for Minorities): a randomized trial of a community health worker intervention to improve diabetic management and control among Bangladeshi adults in NYC. BMC Public Health. 2014 Feb 18;14:177. doi: 10.1186/1471-2458-14-177. PMID 24548534